CLINICAL TRIAL: NCT00888225
Title: Chronic Lateral Epicondylitis. A Randomized Controlled Clinical Trial of Two Physical Training Concepts With Special Reference to Etiology and Treatment Effect
Brief Title: Tennis Elbow Trial
Acronym: Epi-X
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: The Swedish Research Council (Other Government); Amersham Foundation (Unknown); Uppsala County Council, Sweden (Other Government)
Responsible Party: Kurt Svärdsudd, professor, section head, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VR K2005
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Last update posted 2009-04-27 (Estimated); Status verified 2009-04

CONDITIONS: Lateral Epicondylitis
Keywords: Tennis elbow; Epicondylitis; Pain; Muscle strength; Quality of life; RCT; Tendinitis; Chronic tennis elbow
MeSH Terms: conditions — Tennis Elbow; Pain; Tendinopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eccentric exercise (Experimental): Group exposed to eccentric exercise treatment
  Interventions: Procedure: Eccentric exercise
- Concentric exercise (Active Comparator): Group exposed to concentric exercise treatment
  Interventions: Procedure: Concentric exercise

INTERVENTIONS:
Procedure: Eccentric exercise — Eccentric exercise treatment performed at home with three sets of 15 repetitions daily
  Arms: Eccentric exercise
Procedure: Concentric exercise — Concentric exercise treatment at home with three sets of 15 repetitions daily
  Arms: Concentric exercise

SUMMARY:
Epi-X is a multicentered randomized controlled clinical trial of chronic lateral epicondylitis with parallel group design and two phases. In the first phase physical exercise treatment is given in the intervention group and expectance in the reference group. In phase 2 eccentric exercise versus concentric is tested.

DETAILED DESCRIPTION:
Chronic lateral epicondylitis is defined as the presence of a "tennis elbow" for more than 3 months. It is a common condition in the general population and often results in long-term sick-leave. The etiology is unknown. A large number of treatments have been tried but none is generally accepted. However, in Achilles tendinitis a new treatment has been shown effective. It consists of eccentric exercise, i.e. work during stretching rather than shortening of the muscle (concentric exercise). The latter is currently the most common treatment method.

This project is a randomised controlled clinical trial of eccentric versus concentric exercise in 205 patients with chronic lateral epicondylitis. Pain and muscle strength were recorded at start of treatment and after 1,2,3,6 and 12 months. Activities of daily life (ADL) and well-being were recorded at start of treatment and after 3, 6 and 12 months. In addition, blood specimens for a number of neural peptides have been sampled. Moreover, the involvement of the peripheral nervous system in the elbow area has been examined in a subsample of patients. A biopsy from 20 patients per treatment group and from 20 healthy subjects, and a positron emission tomography (PET) scan of 23 patients were performed to allow qualitative and quantitative examination of neural fibres, peptides and receptors. The health economy of the two treatments will be investigated using data from this project and from available registers.

ELIGIBILITY:
Inclusion Criteria:

* Verified tennis elbow for more than three months
* Age 20-75 years
* Informed consent

Exclusion Criteria:

* Inability to understand or follow instructions
* Inability to read or fill in questionnaires
* Inability to participate at measurement sessions
* Supinator syndrome
* Compartment syndrome of anconeus muscle
* Rhizopathy of arm
* Inflammatory joint or soft tissue disease including fibromyalgia
* Previous surgery because of tennis elbow

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2003-10; Primary Completion 2008-01 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Pain during dynamic and static muscle load | Month 0, 1, 2, 3, 6, 12

SECONDARY OUTCOMES:
Muscle strength and function | Month 0, 1, 2, 3, 6, 12

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Svärdsudd, MD, PhD, Principal Investigator — Uppsala University
Locations (2):
- Sweden (2):
  - Linköping University, Linköping
  - Uppsala University, Dept of Public Health and Caring Sciences, Family Medicine and Clinical Epidemiology Section, Uppsala

REFERENCES:
- [Derived] Peterson M, Svardsudd K, Appel L, Engler H, Aarnio M, Gordh T, Langstrom B, Sorensen J. PET-scan shows peripherally increased neurokinin 1 receptor availability in chronic tennis elbow: visualizing neurogenic inflammation? PLoS One. 2013 Oct 14;8(10):e75859. doi: 10.1371/journal.pone.0075859. eCollection 2013. PMID 24155873
- [Derived] Peterson M, Butler S, Eriksson M, Svardsudd K. A randomized controlled trial of exercise versus wait-list in chronic tennis elbow (lateral epicondylosis). Ups J Med Sci. 2011 Nov;116(4):269-79. doi: 10.3109/03009734.2011.600476. PMID 22066975
- See also: Uppsala University, Department of Public Health and Caring Sciences, Family Medicine and Clinical Epidemiology Section, Sweden — http://www.pubcare.uu.se